CLINICAL TRIAL: NCT01614379
Title: Non-enhanced Magnetic Resonance Angiography of Diabetic Ischemic Lower Limbs
Status: Withdrawn | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Michael Vaeggemose, Research Assistant, Aarhus University Hospital
Other Study IDs: 2012-33818
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 1; Ischemia; Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Ischemia; Foot Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample less then 250ml to determine Hba1c (blood glucose level).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy control subject: 10 healthy control subjects for statistical comparison
- Type 1 diabetic patient: 40 type 1 diabetic patients with diabetic foot ulcers.

SUMMARY:
Diabetic foot ulcers often progresses after many years of diabetes where the patients system is so damaged that normal heeling of ulcers cannot happen. The physician at the clinic examines the foot, measuring its circulation and sensitivity. The measures are the blood pressure in comparison between foot and upper arm and oxygen level in the foot. The measurements have a direct connection to the blood circulation, but it doesn't visualize the blood circulation.

Development of MR methods without the use of contrast agents have become so good that images of the blood veins can be used in treatment. This means that the MR images provide important information about the patient vessel wall stiffness and blood circulation without the use of the damaging substances. Hence the physician can perform the MR examination and in comparison with the test performed at the clinic he can make an improved and without risk diagnose. Using MR at a lot earlier stage in the treatment is expected to reduce the number of amputations. This is not only an economic advantage, but also an improvement of the patient quality of life.

The objective of the study is to investigate type 1 diabetics oxygen level, vessel wall stiffness, blood circulation, tissue contribution and blood pressure in the foot with the use of conventional measurements in their treatment and with the added use of MR methods.

This will provide the physician with valuable information of the patient illness and is expected to play an important role in the prevention of diabetic foot ulcers. We expect that MR research leads to a much improved prevention and treatment of aggressive and destructive diabetic foot ulcers. This will increase the general quality of life and reduce the large number of amputations performed every year.

DETAILED DESCRIPTION:
NON-ENHANCED MAGNETIC RESONANCE ANGIOGRAPHY OF DIABETIC ISCHEMIC LOWER LIMBS

BACKGROUND

Diabetic foot ulcers often progresses after many years of diabetes where the patients system is so damaged that normal heeling of ulcers cannot happen. The patient seeks a doctor and he sends the patient to the ulcer clinic or an ulcer specialist. The physician at the clinic examines the foot, measuring its circulation and sensitivity. The measures are the blood pressure in comparison between foot and upper arm and oxygen level in the foot. The measurements have a direct connection to the blood circulation, but it doesn't visualize the blood circulation.

Visualization of the circulation is often achieved with medical imaging methods such as x-ray and MR. The problem with the current use of these methods is the added use of contrast agent. This is especially a problem with the diabetics who have reduced kidney function, where to this method is poisonous to the kidneys. That is why the methods often are only used right before a scheduled amputation, so the surgeon can plan the amputation.

Development of MR methods without the use of contrast agents have become so good that images of the blood veins can be used in treatment. This means that the MR images provide important information about the patient vessel wall stiffness and blood circulation without the use of the damaging substances. Hence the physician can perform the MR examination and in comparison with the test performed at the clinic he can make an improved and without risk diagnose. Using MR at a lot earlier stage in the treatment is expected to reduce the number of amputations. This is not only an economic advantage, but also an improvement of the patient quality of life.

The use of MR technique will furthermore provide the physician with the possibility to create a 3D model of the foot, with segmentation of the different types of tissue in the foot. This makes a single MR scan provide the physician with important information of the physiology (how the foot works), the placement of the ulcer, shape, depth and tissue contribution.

INVESTIGATOR, SPONSOR AND TRAIL SETTING

Michael Vaeggemose is the investigator and will perform the conventional test at the Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Nørreborgade 44, 8000 Aarhus, Denmark. Furthermore Michael will perform the MR scans at the MR Centre, Aarhus University Hospital, Skejby, 8200 Aarhus N, Denmark.

The blood test which is included in the project will be performed by a laboratory technician at the Department of Endocrinology and Internal Medicine. The test is used to determine blood glucose (the sugar level of the blood) and will be destroyed after the examination. There will not be established a biological bank in this project.

Physician Niels Ejskjaer from the Department of Endocrinology and Internal Medicine is attached to project as responsible physician. Niels Ejskjaer will furthermore work as supervisor of the investigator and is the sponsor of this research project.

OBJECTIVE

The objective of the study is to investigate type 1 diabetics oxygen level, vessel wall stiffness, blood circulation, tissue contribution and blood pressure in the foot with the use of conventional measurements in their treatment and with the added use of MR methods.

METHODS

The study is an investigation of MR methods in the treatment of diabetic foot ulcers. The trial consists of 5 physiological examinations and a blood test. To make sure that all the test subjects (diabetics and healthy controls) receive the same treatment is the test performed by the same investigator, with an exception of the blood test which will be performed by the laboratory technician. The 4 test are known to the diabetic patients from earlier clinical trials performed in relation to the treatment of their ulcers, alas they will have to be performed again. Due to logistics the participants can experience more than one day of trail, since the MR clinical and the Department of Endocrinology and Internal Medicine is not placed in the same part of town.

The blood test is used to determine the subjects' blood glucose (the level of sugar in the blood) and will after use be destroyed. Blood glucose level gives a well-defined measure of diabetes. Therefore it is an important measure in the comparison between the conventional test and the MR imaging. Do the blood glucose levels correlate with the findings of the 5 tests then the results of the statistics are plausible and significant results are accepted.

Tree of the test are made in regard to the pulse in the foot. The pulse is measured several places by placing the finger on one of the blood veins in the foot and then count the number of pulse ripples each minute. This is a very simple measurement but effective in estimating the condition of the circulation in the foot. The trails include a more advanced method to measure the pulse at the ankle, middle foot and in the toes compared with the pressure in the arm give an indication of reduced circulation in the specific areas. The measurements are performed with ultrasound and pressure sensitive sensors placed on the pulsating veins.

The fourth examination measures the oxygen level in the foot. Diabetics with foot ulcers often have reduced oxygen level in the feet, which makes the heeling slow and troublesome. This makes the oxygen levels an important measure which is measured in a device connected to the patient with electrodes. The first 4 measurements are all conventional measurements used and performed in the clinic doing the normal treatment of their ulcers.

The MR measurement is used to determine the anatomy and function of the foot. De different scan sequences makes it possible to visualize blood vessels, tissue contribution, oxygen levels and through data processing vessel wall stiffness. Several of the scan sequences are recorded in synchrony with the heart rhythm. The rhythm is recorded wireless with and ECG device after placing of 3 electrodes. The scan time can vary, due to the subjects different heart rates in practice this means that the MR scans takes from 30 min to 60 min.

STATISTICAL CONSIDERATIONS

Sensitivity and specificity of the MR methods will be evaluated I relationship to the conventional applied methods (pulse and oxygen level measurements) which will be performed at the Department of Endocrinology and Internal Medicine. From a McNemar's test with a significant level of 5% a power calculation were performed giving a needed sample size of 40 type-1 diabetic patients and 10 healthy control subjects. To perform the statistical calculations assumptions of the sensitivity and specificity have been made. Due to the assumptions a pilot study will be performed with 5 diabetic patients showing if the MR method produces enough signal to make the need examination.

VOLUNTEERS

The trails consist of 10 healthy (don't use prescribed medicine) and 40 type-1 diabetic foot ulcer patients. Subjects from both groups are at least 18years old and have received oral and written information regarding the project and afterward given informed consent of participation in the project. Furthermore a requirement of the diabetic foot ulcers is that the ulcer must have a reduced oxygen level.

Subjects will be excluded if they have metal in the body or are scheduled to have an amputation as part of their treatment.

SIDE EFFECTS, RISK AND DISADVANTAGES

Oxygen level and pulse examinations meet the requirements of patient safety and are used in a large number of examinations. There are no known risks in the used methods but should there be an unpleasantness or problems from regarding the participation the patient must contact the investigator at once.

MR scans is also not connected to any known risks and the patients ears will be protected with soundproofing earplugs or headphones to avoid the discomfort in relation to the high sound the scanner makes during the scans. The patient will be placed outside the scanner, with the feet sticking into the scanner, removing the risk of making the patient feel claustrophobic.

The blood test can be connected to slight discomfort and a small risk of developing accumulation of blood and infection at the needle injection site. If any sign of infection (rash, heating, tenderness, swelling) the subject must seek the investigator or the emergency room. Det combined blood loss in connection to the blood test will not exceed 250ml, which is a lot less than a blood donation includes.

The blood test is analysed and destroyed after. A biobank will not be established in this project.

ECONOMIC CONDITIONS

Expenses in connection to the project are covered by the involved departments. The researchers have no economic conflict of interest in the project. Transport expenses in connection to oral information and examination is refunded in regard to the guidelines used at the departments. In regard to national guidelines the subjects will be paid compensation for their partition in the project.

PUBLICATION OF RESULTS

The results will be published in a recognized international paper regardless of the results are positive, negative or if the method is not good enough to determine a statistical significant difference.

Do the subjects wish information about the project results they can inform the investigator and he will send the information to the interested subjects.

NATIONAL ETHICAL COMMITTEE REVIEW

The project is reported and approved by the Danish Data Protection Agency (nr. 2007-58-0010), Danish National Committee on Health Research Ethics (nr. 2012-33818) and the department legislations.

VOLUNTEER RECRUITMENT

Diabetic subjects with foot ulcers will be asked of interest to participate in the study, when visiting the clinic in connection to their regular treatment at the clinic. Staff physician Niels Ejskjaer is treating a large part of the patients and will after their visit at the clinic ask the patients of participation, with stretch on that it's voluntary and it has not effect of their regular treatment. If a patient agree to participate he/she will receive information of the project and information of participation in research projects (Forsøgspersonernes rettigheder i et sundhedsvidenskabeligt forskningsprojekt) written by the Danish National Committee on Health Research Ethics.

Latest a week after receiving the information investigator Michael Vaeggemose will contact the subject and ask if he/she still wishes to participate and would like to hear more about the aspects of the project. Furthermore the patient will be invited to a personal conversation with the possibility to have a trusted friend in the room that can help the patient in the choice of participating in the project. The healthy control subjects will be recruited from posters calling for participants to contact the investigator on phone or mail. The posters will have information about the project but information on the phone and invitation to a personal conversation with a trusted friend will be offered, as it is to the diabetic patients. The conversations (diabetic and control) will be held undisturbed in one of the department rooms. At the conversations it will be stretched that participating is volunteer and as a volunteer you can chose to stop you participation at any point in the project, without it having any effect on their following treatment. During the conversation the patient is given the written consent document which must be signed before the trails can begin. The patient has a week to evaluate the project from this point and will then receive a call from the investigator regarding the final decision of participating in the project.

ELIGIBILITY:
Inclusion Criteria (diabetic group):

* Type 1 diabetic patient with ischemia in the lower extremities determined from conventional clinical measurements (palpable foot pressure, ankle-brachial index, transcutaneous oxygen level, toe pressure).
* Diabetic foot ulcer with a Wagner score of 0-2.

Inclusion Criteria (healthy control group):

* Do not use prescription drugs.
* BMI is between 20 and 30.

Exclusion Criteria:

* If subject does not apply to the MR safety rules.
* Less then 18 years old.
* Has a planed amputation of a lower extremity as part of treatment.
* Diabetic foot ulcer with a Wagner score of 3-5.
* Internal insulin pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic subjects with foot ulcers will be asked of interest to participate in the study, when visiting the clinic in connection to their regular treatment at the clinic. Staff physician Niels Ejskjaer is treating a large part of the patients and will after their visit at the clinic ask the patients of participation, with stretch on that it's voluntary and it has not effect of their regular treatment.
  The healthy control subjects will be recruited from posters calling for participants to contact the investigator on phone or mail. The posters will have information about the project but information on the phone and invitation to a personal conversation with a trusted friend will be offered, as it is to the diabetic patients.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaeggemose, MSc, Principal Investigator — Department of Endocrinology and Internal Medicine, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Endocrinology, Aarhus, Denmark
  - MR Centre, Aarhus, Denmark